CLINICAL TRIAL: NCT03903757
Title: Network-based Epigenome-Wide associaTion Study in Obesity precisioN Medicine: NEWTON Clinical Trial
Brief Title: Network Medicine, Epigenetics and Obesity
Acronym: NEWTON
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Giuditta Benincasa, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: PRIN2017F8ZB89
Record Dates: First submitted 2019-03-31; First posted 2019-04-04 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Obesity; Type2 Diabetes
Keywords: Epigenetics; Network medicine; Personalized therapy
MeSH Terms: conditions — Obesity | interventions — Epigenome; Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subcutaneous adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese subjects with and without T2D
  Interventions: Other: DNA methylome and total RNA sequencing
- control subjects
  Interventions: Other: DNA methylome and total RNA sequencing

INTERVENTIONS:
Other: DNA methylome and total RNA sequencing — Epigenomics tools combined with bioinformatic analysis to correlate putative useful clinical biomarkers with clinical features

SUMMARY:
The prevalence of obesity is increasing and affects more than 650 million people of all ages to become one of the foremost global health threats. Obesity is a complex syndrome that can seriously impair health through a broad range of complications such as cardiovascular disease, type 1 and 2 diabetes (T1D and T2D), cancer, musculoskeletal disorders, psychosocial imbalances, and reduced quality of life, and impacts the treatment of other conditions. Weight reduction has been shown to have a positive effect on these co-morbidities and may increase the effectiveness of treatments specific for other co-morbidities. Lifestyle modification is an integral part of the weight management journey, but is often insufficient on its own, and can be complimented by pharmacological and surgical add-on treatments to achieve greater and more sustainable weight loss, as appropriate. It is likely that there are subgroups of patients that are more suited to certain types of treatment and results risk dilution of perceived efficacy unless these groups are identified and treatment is personalised. The aim of this project is to identify pathophysiologically and clinically meaningful subgroups of obesity by performing Next Generation Sequencing (NGS) approaches and network based algorithm that will allow the optimisation of prevention and treatment of obesity and its complications.

DETAILED DESCRIPTION:
Population study will be recruited at the Clinical Department of Internal Medicine and Specialistics, Department of Advanced Clinical and Surgical Sciences belonging to University of Campania "Luigi Vanvitelli". This study will be performed according to the principles outlined in the Helsinki Declaration. Subcutaneous adipose tissues located in the surgical incision will be withdrawn without the use of surgical devices in order to avoid the degradation of the biological sample from 50 obese subjects (25 obese subjects with Type 2 Diabetes vs 25 obese subjects without Type 2 Diabetes) undergoing bariatric surgery. As controls (n=50) we will recruit subcutaneous adipose tissues from patients without a clinical history of cardiovascular or dysmetabolic diseases undergoing to surgery for stress inguinal hernia. Clinical and demographic characteristics of the study population will be available from datasets generated by physicians.

From tissue samples the genomic DNA and the total RNA will be extracted. Genomic DNA will be extracted by using DNeasy Blood & Tissue kit (QIAGEN), according to manufacturer protocol. Pooled DNA samples consisting of equal quantities of DNA (2 µg) from cases and controls will be shipped to Genomix4Life Genomics and Bioinformatics Service, to perform a global DNA methylation analysis. For this aim, it will be used the Human Methylation 27K BeadChip platform by using Bisulfite conversion technology (BBRS-Seq). Total RNA will be extracted from tissues using RNeasy Mini Kit (QIAGEN) according to manufacturer protocol. The cDNA library preparation will be performed starting from 4 ug of total RNA by using Illumina TruSeq Libraries and then sequenced at high coverage on the Illumina HiSeq 2500 NGS platform. Nucleic acid concentrations and quality control from Genomix4Life will be assessed by using Nanodrop spectrophotometer (Thermo Fisher Scientific) and Qubit assay (Thermo Fisher Scientific) and TapeStation 4200 (Agilent). The weighted human DNA methylation PPI network (WMPN) will be construct to obtain a obesity interactome in both subgroups (obese and obese with T2D vs controls) based on differentially methylated genes in order to identify putative useful diagnostic biomarkers. The TargetScan algorithm , by searching the conserved seed pairing regions in the 3' untraslated regions (UTR) of genes based on whole genome alignment, will be used to robustly predict miRNA-target gene pairs from the same study population.

ELIGIBILITY:
Inclusion Criteria:

* Meets the current American Diabetes Association guideline for diagnosis of diabetes (Diabetic group) and obesity
* Must be willing and able to comply with study requirements
* Must indicate their understanding of the study and willingness to participate by signing an appropriate informed consent form

Exclusion Criteria:

* History of cancer
* Malignancy disorders
* Active infections
* Chronic or immune-mediated diseases
* Primary disease requiring surgical intervention
* Unable to comply with the complication screening
* Less than 18 y of age
* Pregnant or are planning to become pregnant during the duration of the investigation
* Life expectancy <12 m
* Currently participating in any other clinical investigation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subcutaneous adipose tissues located in the surgical incision will be withdrawn without the use of surgical devices in order to avoid the degradation of the biological sample from 50 obese subjects (25 obese subjects with Type 2 Diabetes vs 25 obese subjects without Type 2 Diabetes) undergoing bariatric surgery. As controls (n=50) we will recruit subcutaneous adipose tissues from patients without a clinical history of cardiovascular or dysmetabolic diseases undergoing to surgery for stress inguinal hernia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
DNA methylation pattern in adipose tissues | 3 months
  Using Methylation 27K BeadChip platform based on Bisulfite conversion technology, DNA methylation profile in adipose tissues of 25 preselected obese subject and 25 obese subjects respect with controls (n=50) will be performed.
Bioinformatics analysis to predict putative novel candidate genes underlying obesity phenotype | 6 months
  The network-based algorithm "Weighted Human DNA methylation PPI network (WMPN)" will be applied to methylome data in order to obtain a disease module containing the crucial differentially methylated genes both in obese patients and obese patients with T2D compared to controls.
RNA sequencing analysisin adipose tissues | 3 months
  RNA sequencing analysis by using Illumina HiSeq2000 Next Generatin Sequencing (NGS) platform will be performed for identifying differentially expressed micro-RNA and mRNA target both in obese patients and obese patients with T2D compared to controls.

SECONDARY OUTCOMES:
ROC curves analysis to evaluate putative DNA methylation/microRNA interactions | 12 months
  ROC curves analysis to evaluate putative DNA methylation/microRNA interactions as diagnostic biomarkers to discriminate obesity subgroups.
Linear regression analysis and BMI (Kg/m2). | 12 months
  Linear regression to correlate epigenetic biomarkers with BMI (Kg/m2) in different soubgroups.
Linear regression to correlate epigenetic biomarkers with proinflammatory cytokines | 12 months
  Linear regression to correlate epigenetic biomarkers with proinflammatory cytokines (TNF-α,IL-6, PCR) levels in different soubgroups.
Linear regression to correlate epigenetic biomarkers with HOMA index | 12 months
  Linear regression to correlate epigenetic biomarkers with clinical variables, such as HOMA index glycemia(mmol/L) x insulinemia (mUI/L)/ 22.5, in different soubgroups.

IPD SHARING:
Plan to Share IPD: No